CLINICAL TRIAL: NCT04840147
Title: A Randomized, Controlled, Comparative, Single-blinded, Multi-center Study Evaluating JointRep® and Microfracture in Repair of Focal Articular Cartilage Lesions on the Femoral Condyle or Trochlea, The JMAC Trial.
Brief Title: A Comparison of JointRep® and Microfracture in Repair of Cartilage Lesions on the Femoral Condyle or Trochlea,
Acronym: JMAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oligo Medic Pty Ltd (Industry)
Collaborators: Mobius Medical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JR001PMAUS01-2020
Record Dates: First submitted 2021-03-23; First posted 2021-04-09 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Chondral Defect; Articular Cartilage Defect; Articular Cartilage Disorder of Knee
Keywords: Bone Marrow Stimulation; Microfracture; Matrix Augmented Bone Marrow Stimulation; Chitosan
MeSH Terms: conditions — Fractures, Stress | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): JointRep® plus microfracture
  Interventions: Device: JointRep®; Procedure: Microfracture
- Control (Other): Microfracture alone
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Device: JointRep® — JointRep® is a medical device based on a thermogel polymer (Chitosan) for the treatment of chondral lesions, which consists of an injectable aqueous composition that forms a solid and sticky hydrogel in situ within cartilage defect(s). JointRep® is composed of an injectable thermo-gelling aqueous composition. It is used in conjunction with a Bone Marrow Stimulation type of procedure like Microfracture.
  Arms: Intervention
Procedure: Microfracture — Microfracture is a bone marrow stimulation type of procedure where after debridement of the damaged chondral tissue within the lesion, obtention of stable vertical margins and curettage of the entire calcified layer, multiple holes are created with a variety of instruments (awls, picks, microdills, nanofracture) to establish a communication with the subchondral bone to create a blood clot to elicit the natural healing process
  Other Names: Bone Marrow Stimulation

SUMMARY:
The aim of the study is to compare whether JointRep® plus microfracture is more effective than microfracture alone when treating symptomatic focal articular cartilage lesions in the knee (femoral condyles or trochlea).

DETAILED DESCRIPTION:
The aim of the JMAC study, an international multicenter Randomized Controlled Trial, is to assess the effectiveness and safety of JointRep®, a second-generation chitosan-based hydrogel for cartilage repair. A total of 185 subjects will be randomized 2:1 to either Microfracture plus JointRep® or Microfracture alone. The follow up will be at 24 months, with a planned interim analysis at 12 months. The primary endpoint is an objectively measured structural one (quantity of new cartilaginous tissue, assessing the percentage of fill) and it will be blindly assessed using a quantitative MRI at 12 and 24 months. Two of the secondary endpoints are also structurally based and blindly measured: quality of the new tissue, quantifying the T2 (which measures the Collagen 2 content and orientation as well as degree of hydration); the upper and lower half of the new tissue T2 measurement will depict the degree of stratification of the new cartilaginous tissue. A semiquantitative MOCART-2 blinded analysis will also be carried out. The clinical outcomes will be measured using KOOS and Tegner, as well as a VAS and an EQ-5 questionnaire. All the secondary endpoints will be analyzed at the same 12 and 24 months timepoints. In addition, subject safety will be assessed through a record of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18-65 years old
* Have one or two focal articular cartilage lesion(s) (ICRS Grade 3 or 4A) on the femoral condyles or trochlea of the index knee; patellar tracking must be normal if the index lesion(s) is on the trochlea. Individually, a lesion can be between 1-7cm2. If more than one lesion is present, the sum of the two lesions should not exceed 10cm2.
* Within 6 months prior to treatment, have a Magnetic Resonance Imaging (MRI) or arthroscopic confirmation of lesion(s) in the index knee.
* For patients older than 40 y.o, to have a radiological Kellgren and Lawrence (K&L) grading from a standing knee radiograph taken less than 6 months previously, Grade 1 or
* If not, an actual test will be performed as part of the visit 1 procedures.
* Have a clinically stable knee, with no ligament deficiencies (<5mm side-to-side difference on Lachman and varus/valgus stress testing & Grade 0 or 1 on Pivot shift test) and the meniscal rims are intact (a maximum of 50% resection is allowed)
* Be able to give voluntary, written informed consent to participate and have signed an Informed Consent Form specific to this study
* VAS pain great than or equal to 4 in the last week.
* Be willing and able to comply with all study procedures including all preoperative, post-operative and rehabilitation requirements
* If female and of child-bearing potential, must report double-barrier, contraceptive use (e.g. use of birth-control pill and condom) for at least 2 months prior to treatment and in the 12 months following treatment.
* If female and of child-bearing potential, have a negative pregnancy test prior to the surgical procedure and no intention of becoming pregnant in the 12 months following treatment.

Exclusion Criteria:

* Have a Body Mass Index (BMI) >35kg/m2
* Have more than two lesions (ICRS grade 3 or 4A) on any surface in the index knee
* Have "kissing" or opposing lesion(s) (ICRS grade 3 or 4A) of the condyle, tibia or patella in the index knee; additional linear lesions which bear Grade 3 or 4 characteristics may be acceptable if they are determined by the Investigator to be incidental, not clinically relevant, and consistent with the subject demographic
* Have malalignment of >5 degrees varus or valgus in the index knee based on standard AP x-rays requiring an osteotomy
* Have had any surgical treatment for cartilage repair in the index knee within 1 year prior to treatment
* Have had intra-articular injections within 3 months in the index knee
* Have a diagnosis of a concomitant knee injury which may confound assessment of the index knee (e.g., important meniscal injury)
* Have significant pain emanating from other lower body joints in the ipsilateral (hip, ankle) or contralateral (hip, knee, ankle) limb.
* Have known allergies to shellfish
* Have a known history of crystalloid or inflammatory arthropathy
* Have any condition that is unrelated to the index knee and significantly impairs walking ability (e.g., spinal stenosis, sciatica)
* Have advanced musculoskeletal disease
* Have active coagulation disorders
* Are currently using antibiotics
* Are participating concurrently in another clinical investigation, or have participated in a clinical investigation within the last 90 days, or intend to participate in another clinical investigation during the course of the study
* Are currently abusing drugs or alcohol or have a history of the same within the last 12 months
* Have any mental or psychological disorder that would impair their ability to complete the study questionnaires
* Are currently breastfeeding or planning to breastfeed any time during the course of the study
* Are currently a prisoner
* Have significant comorbidities or conditions associated with high-risk for surgical or anesthetic survival (e.g., renal failure, peripheral vascular disease, unstable cardiac disease, poorly controlled diabetes, immunosuppression, etc.)
* Have any medical condition or other circumstances, in the judgment of the investigator, that might interfere with the ability to return for follow-up visits, including any systemic illness, neuromuscular, neurosensory, or musculoskeletal deficiency that would render the subject unable to perform appropriate post-operative rehabilitation
* Have any condition which, in the judgment of the Investigator, would preclude adequate evaluation of the device's safety and performance

Intra-operative Exclusion Criteria:

Subjects who meet any of the following intra-operative screening criteria will be excluded from participation in this study:

* Have lesion(s) in the index knee that are not contained (intact shoulders) and/or exceed 7 cm² in total size after debridement for a single lesion and 10cm2 for more than one lesion, if within the same condyle or the trochlea. If only a single lesion suitable to be included is identified, it might be between 1-7cm2.
* Minor concomitant procedures are allowed such as, but not limited to:

  1. Removal of loose bodies
  2. Plica excision
  3. Minor synovial removing
  4. Minor chondroplasty (debridement)
  5. Lysis of adhesions
  6. Meniscal trimming/suturing which respects the exclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Lesion fill. | 24-months post procedure.
  Percentage of lesion fill measured by 3D quantitative Magnetic Resonance Imaging (qMRI).

SECONDARY OUTCOMES:
Visual Analogue Scale. | Baseline and then at 3-months, 6-months, 12-months and 24-months post procedure.
  Pain score in treated knee using the visual analogue scale from 0(no pain) to 10 (worst pain imaginable) .
T2 scores. | 12 and 24-months post procedure.
  Difference in quantitative T2 scores between investigational subjects and control subjects measured by qMRI.
Treatment failure. | 24-months post procedure.
  Proportion of subjects who do not experience a treatment failure and achieve ≥80% lesion fill (success rate).
Knee Injury and Osteoarthritis Outcome Score (KOOS). | 6 and 12 and 24-months post procedure.
  Knee Injury and Osteoarthritis Outcome Score (pain, function, symptoms, sports/recreation and quality of life). 100 indicates no problems and 0 indicates extreme problems.
Tegner Activity Scale | 6 and 12 and 24-months post procedure.
  Tegner activity scale provides a level of activity and is scored between 0 and 10. Level 0 is the worst activity level and Level 10 is the best activity level.
Magnetic Resonance Observation of Cartilage Repair Tissue 2.0 (MOCART-2) score. | 6 and 12 and 24-months post procedure.
  MOCART-2 score ranges form 0 (worst outcome) to 100 (best outcome) .
Euro Quality of Life-5D (EQ-5D) instrument for measuring quality of life. | 6 and 12 and 24-months post procedure.
  EuroQol-5D (EQ-5D) instrument for measuring quality of life has two parts. The first assesses health in five parts (mobility, self-care, usual activity, pain/discomfort, anxiety depression) with each scored form 1 (best outcome) to 5 (worst outcome). The second part consists of a visual analogue scale rating perceived health form 0 (the worst imaginable health) to 100 (the best imaginable health).
Safety as Adverse Events related to the procedure | Baseline to 24-months post procedure.
  Evaluation of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Caldwell, MBBS, FRACS, Principal Investigator — Lingard Private Hospital
Locations (8):
- Australia (7):
  - Canberra Orthopaedics and Sports Medicine, Deakin, Australian Capital Territory
  - Sydney Knee Specialists, Kogarah, New South Wales
  - Lingard Private Hospital, Newcastle, New South Wales
  - Orthosports, Randwick, New South Wales
  - Cairns Orthopaedic Clinic, Parramatta Park, Queensland
  - North Queensland Knee, Pimlico, Queensland
  - Melbourne Orthopedic Group, Melbourne, Victoria
- Dartmouth General Hospital, Dartmouth, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No